CLINICAL TRIAL: NCT03337802
Title: Effect of Mediterranean Diet During Pregnancy on the Onset of Overweight and Obesity at 24 Months in the Offspring
Brief Title: Effect of Mediterranean Diet During Pregnancy on the Onset of Overweight and Obesity in the Offspring
Acronym: PREMEDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 298/16
Record Dates: First submitted 2017-11-02; First posted 2017-11-09 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant women at standard diet (No Intervention): obstetrical and gynecological follow-up
- Pregnant women at mediterranean diet (Experimental): obstetrical and gynecological follow-up + nutritional counseling
  Interventions: Behavioral: mediterranean diet

INTERVENTIONS:
Behavioral: mediterranean diet — The Mediterranean diet (MD) is highly regarded as a healthy balanced diet. It is distinguished by a beneficial fatty acid profile that is rich in both monounsaturated and polyunsaturated fatty acids, high levels of polyphenols and other antioxidants, high intake of fiber and other low glycemic carbohydrates, and relatively greater vegetable than animal protein intake. Specifically, olive oil, assorted fruits, vegetables, cereals, legumes, and nuts; moderate consumption of fish, poultry, and red wine; and a lower intake of dairy products, red meat, processed meat and sweets characterize the traditional MD.
  Arms: Pregnant women at mediterranean diet

SUMMARY:
The first 1,000 days of life, from the conception to 24 months, are crucial to achieve long-term health outcomes and represent a strategic period to intervene under prevention and public health perspective. Nutritional exposures during this critical period of life can influence the future disease susceptibility. Maternal diet during pregnancy has been linked to offspring overweight/obesity risk and it could represent a potential target for overweight/obesity prevention. The Mediterranean Diet (MD) is considered one of the healthiest dietary models, which impacts beneficially the gut microbiome (GM), providing high amounts of fiber, antioxidants polyphenols and vitamins, and a balanced ratio of essential fatty acids (ω6:ω3). Notably, the MD beneficial effects are due to the synergistic and interactive combinations of nutrients, and the modulation of gene expression through epigenetic changes. Unofrtunately, the MD mechanisms during pregnancy in the prevention of childhood overweight/obesity are not yet fully known.

DETAILED DESCRIPTION:
The PREMEDI study has been designed to evaluate the effects of Mediterranean Diet during pregnancy on the occurrence of overweight/obesity at 24 months in the offspring.

ELIGIBILITY:
Inclusion Criteria:

* women
* caucasian ethnicity
* aged between 20 and 35 years

Exclusion Criteria:

* proven presence of infections during pregnancy and at delivery,
* twin pregnancy,
* ongoing malignancies,
* major gastrointestinal tract malformations,
* immunodeficiencies,
* diabetes and other chronic diseases at each organ or apparatus level,
* chronic intestinal inflammatory diseases,
* gastrointestinal function disorders,
* celiac disease;
* history of abdominal surgery with intestinal resection,
* neuropsychiatric disorders,
* central nervous system disorders,
* vegan diet.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
The effects of Mediterranean Diet in pregnancy on the occurrence of overweight/obesity at 24 months in the offspring | After 24 months from the delivery
  The children body growth indices are evaluated at 24 months

SECONDARY OUTCOMES:
The effect of Mediterranean Diet pregnancy on the composition of maternal gut microbiota through analysis of gut microbiota composition. | after 9 months (at the end of the pregnancy)
  Fecal bacteria DNA will be extracted using standard technique outlined by the Earth Microbiome Project. 16S V4-region amplicon libraries will be produced using previously described primers and sequenced using the IlluminaMiSeqplatform (150bpx2). Bacterial load will be determined by qPCR using a standard curve derived from a plasmid containing a single copy of the 16S rRNAencoding gene. Sequence data has been deposited in MG RAST under accession numbers 4571868.3-4571924.3 and project number 10023. Paired end reads will be quality trimmed and processed for OTU (operational taxonomic unit) clustering using UPARSE pipeline, set at 0.97% identity cutoff. Taxonomic status will be assigned to the high quality (<1% incorrect bases) candidate OTUs using the "parallel_assign_taxonomy_rdp.py" script of QIIME software. Multiple sequence alignment and phylogenetic reconstruction will be performed using PyNast and FastTree.
The effect of Mediterranean diet in pregnancy on the production of short chain fatty acids (butyrate and propionate) in the intestinal tract. | after 9 months (at the end of the pregnancy)
  Fecal SCFAs concentration Frozen feces weighing 1g will be diluted with saline solution, vortexed, and centrifuged. Supernatants will be filtered and stored at -20°C until analysis. Frozen fecal extracts will be acidified and extracted in duplicate. A quantity of the pooled extract containing acidified butyrate, propionate or acetate will be transferred into a 2ml glass vial and loaded onto an Agilent Technologies 7890 gas chromatograph (GC) system. Detection will be achieved using a flame ionization detector. Peaks will be identified using a mixed external standard and quantified by peak height/internal standard ratio. To examine whether fecal butyrate levels correlates with bacterial diversity (Shannon diversity index) and evenness (Pielou's evenness index) and abundance patterns across multiple groups we will calculate the Spearman correlation using the cor.test function implemented in R (http://www.r-project.org/
The adherence to Mediterranean Diet in the enrolled women | from 0 to 9 months (at the end of pregnancy)
  Women Mediterranean Diet adherence score is evaluated through the "Med Diet Score"
The effect of dietary counseling on dietary habits | from 0 to 9 months (at the end of pregnancy)
  The diet composition in macro- and micronutrients is evaluated
The effect of Mediterranean diet in pregnancy on the maternal weight gain and complications | from 0 to 9 months (at the end of pregnancy)
  To evaluate the effect of Mediterranean diet in pregnancy on the maternal weight gain and complications (gestational hypertension, infections, gestational diabetes, preeclampsia, use of cesarean)
The effect of Mediterranean diet in pregnancy on perinatal and fetal complications | from 0 to 9 months (at the end of pregnancy)
  Perinatal and fetal complications occurrence are evaluated
The effect of Mediterranean Diet in pregnancy on the duration of breastfeeding and the composition of breast milk | from 0 to 4 months lactation
  The effect of Mediterranean Diet in pregnancy on the duration of breastfeeding and the composition of breast milk (short chain fatty acids, bacterial DNA, adipocytokines.
The effect of Mediterranean Diet on the occurrence of allergies and use of antibiotics in the first 2 years of life. | Every 6 months from offspring birth to 2 years
  The occurrence of allergies and the use of antibiotics in the first 2 years of life are evaluated
The effect of Mediterranean Diet on the epigenetic modulation of genes involved in the regulation of immune system and metabolic pathways in the offspring | At delivery
  The evaluation of the effect of Mediterranean Diet during pregnancy on the epigenetic modulation of genes involved in the immune system and metabolic pathways in the offspring through the cord blood epigenome-wide association study

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Berni Canani, Principal Investigator — Department of Traslational Medical Science, University of Naples Federico II
Locations (1):
- University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coppola S, Paparo L, Bedogni G, Nocerino R, Costabile D, Cuomo M, Chiariotti L, Carucci L, Agangi A, Napolitano M, Messina F, Passariello A, Berni Canani R. Effects of Mediterranean diet during pregnancy on the onset of overweight or obesity in the offspring: a randomized trial. Int J Obes (Lond). 2025 Jan;49(1):101-108. doi: 10.1038/s41366-024-01626-z. Epub 2024 Sep 18. PMID 39289583